CLINICAL TRIAL: NCT01390116
Title: The Effect of Aged Garlic Extract Supplementation on Immune System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Wakunaga Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AGE-84403
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Improvement in Immune Cell Function in Healthy Humans
Keywords: gamma delta T cell; natural killer cell; proliferation; cytokine secretion; Improvement in immune cell function in healthy humans
MeSH Terms: interventions — kyolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator): looks like and is given in the same way as the experimental treatment but contains no active ingredient
  Interventions: Dietary Supplement: Aged garlic extract
- AGE (Experimental): Encapsulated aged garlic extract, 4 capsules per day, 2.56 g/day
  Interventions: Dietary Supplement: AGE

INTERVENTIONS:
Dietary Supplement: Aged garlic extract — 2 aged garlic extract capsules taken twice daily
  Other Names: AGE
  Arms: Sugar pill
Dietary Supplement: AGE — encapsulated aged garlic extract, 4 capsules per day, 2.56g/day
  Other Names: Kyolic
  Arms: AGE

SUMMARY:
The purpose of this study is to determine whether consuming capsules of aged garlic extract is effective in enhancing function of NK and/or γδ T cell resulting in fewer cold and flu symptoms.

DETAILED DESCRIPTION:
A non-therapeutic intervention study is described. The Aged Garlic Extract (AGE) supplement (and placebo) intervention occurs over a total of 90 days between mid-January to March. The CDC indicates that this is the cold and flu season (http://www.cdc.gov/flu/weekly/fluactivity.htm ). Blood is taken at baseline and at 45 days, 2 hours after they have taken their capsule. Capsule consumption will continue for a total of 90 days in order to continue monitoring cold and flu symptoms. Subjects will be given a diary to keep a record of their cold and flu symptoms. Peripheral blood mononuclear cells are isolated from the blood draw and used fresh, cultured in autologous serum for 24 hours or cultured in autologous serum for 10 days. Freshly isolated cells will be used for glutathione analysis, for protection against induced DNA strand breaks, and for γδ T cell and NK cell numbers. The supernatant of 24 hour cultures will be used for cytokine determination, specifically, interferon-g, tumor necrosis factor-a and IL-12. Cells cultured for 10 days will be used to determine the rate of proliferation. If cells have been primed by AGE, we expect the AGE cells to proliferate to a greater extent and have greater cytokine secretion compared to placebo.

If AGE enhances the function of one or both of these cell types (NK or γδ T cell), then it is possible that there will be fewer cold and flu symptoms in the group consuming the supplement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female
* Between the ages of 21 and 50
* BMI between 18 and 35

Exclusion Criteria:

* High blood pressure defined as 140/90
* Ongoing or chronic illness or infection
* On hypertensive medication, immunosuppressive drugs, antibiotics, or chronic use of NSAIDS
* Taking dietary supplements other than those with "normal" levels of vitamins and minerals
* Consumes more than 2 glasses of alcoholic beverages per day

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Physiological modifications to immune cell function | 45 days
  The ability of the natural killer and/or γδ T cells to proliferate when cultured ex vivo.

SECONDARY OUTCOMES:
Cold and flu symptoms | 90 days
  Incidence and severity of cold and flu symptoms, total and individual. Other signs of severity, for example, visits to doctor or health clinic, reduction in daily activities, medications prescribed or purchased OTC.
Cold and flu symptoms | 90 days
  Incidence and severity of cold and flu symptoms, total and individual. Other signs of severity, for example, visits to doctor or health clinic, reduction in daily activities, medications prescribed or purchased Over the Counter (OTC).

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Percival, PhD, Principal Investigator — University of Florida
Locations (1):
- 449 Food Science and Human Nutrition Department, Gainesville, Florida, United States

REFERENCES:
- [Derived] Percival SS. Aged Garlic Extract Modifies Human Immunity. J Nutr. 2016 Feb;146(2):433S-436S. doi: 10.3945/jn.115.210427. Epub 2016 Jan 13. PMID 26764332
- [Derived] Nantz MP, Rowe CA, Muller CE, Creasy RA, Stanilka JM, Percival SS. Supplementation with aged garlic extract improves both NK and gammadelta-T cell function and reduces the severity of cold and flu symptoms: a randomized, double-blind, placebo-controlled nutrition intervention. Clin Nutr. 2012 Jun;31(3):337-44. doi: 10.1016/j.clnu.2011.11.019. Epub 2012 Jan 24. PMID 22280901